CLINICAL TRIAL: NCT02526797
Title: Multiparametric MRI in Men With Prostate Cancer Undergoing Active Surveillance
Status: Enrolling by invitation | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Lars Boesen, MD, PhD, Herlev Hospital
Other Study IDs: HEH-2015-058
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Neoplasms
Keywords: prostate biopsy; prostate cancer; Magnetic resonance imaging; Neoplasm staging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate whether multiparametric MRI (mp-MRI) in patients with low-risk prostate cancer can improve the selection of patients suitable for Active Surveillance and have a relevance in the ongoing monitoring.

DETAILED DESCRIPTION:
Men with localized prostate cancer (PCa) with small tumor burden may be followed on active surveillance (AS) rather than active treatment. AS is an attempt to avoid over-treatment of PCa, which is estimated to be insignificant at the time of diagnosis, and therefore unlikely to affect patient morbidity and mortality. AS include close monitoring with PSA measurement (blood test), digital rectal exploration (DRE) and trans-rectal ultrasound-guided prostate biopsy (TRUS-bx) at regular intervals, so that active treatment can be initiated if the cancer becomes more aggressive. It is crucial that patients undergoing AS are staged correctly, to avoid underestimating more aggressive disease and patients mistakenly are enrolled into AS instead of active treatment.

Previously, a PhD study conducted at Herlev Hospital revealed that multiparametric MRI (mp-MRI) of the prostate can improve the detection and staging of PCa and may add additional information about tumor aggressiveness compared to the traditional methods DRE and TRUS-bx. Mp-MRI at the inclusion of AS may detect missed significant tumors and potential areas of higher aggressiveness than detected by the traditional biopsies. Additional targeted biopsies from these suspicious areas can then be performed with a re-evaluation of the treatment plan, if more advanced disease is identified. Conversely, mp-MRI has a high negative predicted value for significant disease and can be used to rule out significant PCa, reassuring patients and physicians to go on with AS. Mp-MRI has been used at the Urology Department, Herlev Hospital, since 2013 in the diagnosis of PCa and in the evaluation of patients undergoing AS. The main objective of this study is to retrospectively investigate, whether mp-MRI can improve the selection of patients suitable for Active Surveillance and have a relevance in the ongoing monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low risk localized prostate cancer enrolled in active surveillance

Exclusion Criteria:

* Metastatic prostate cancer
* No mp-MRI data present
* Prostate cancer treatment
* Known allergic reaction to Gadolinium-based MRI contrast agent
* Prostate biopsy during the last 21 days
* Impaired renal function with GFR < 30 ml / min
* pacemaker
* Magnetic metal residues in the body
* Claustrophobia
* Psychiatric disorders
* Age under 18 years

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with newly diagnosed low-risk prostate cancer enrolled in active surveillance at Dept. of Urology, Herlev University Hospital, from Januar 2013 to June 2015, who have had an mp-MRI of the prostate in their diagnostic follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the treatment planning from active surveillance to active treatment based on mp-MRI | 3 months
  Observe changes in the detection-rate of significant prostate cancer using mp-MRI and mp-MRI targeted biopsies in men with newly diagnosed low risk prostate cancer enrolled i active surveillance. Mp-MRI is performed approximately 2½ month after the initial prostate biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Boesen, MD, PhD, Principal Investigator — Department of Urology, Herlev University Hospital Herlev, Herlev, Denmark, 2730
Locations (1):
- Department of Urology, Herlev University Hospital Herlev, Herlev, Denmark